CLINICAL TRIAL: NCT01599546
Title: Reading in Preterm and Full-term Children: Neural Basis and Prediction
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heidi M. Feldman, MD, PhD, Stanford University
Other Study IDs: IRB-22233
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Premature Birth; Basic Learning Problem in Reading; Child
Keywords: Preterm; Full term; Reading; Dyslexia; Brain; Diffusion tensor imaging
MeSH Terms: conditions — Premature Birth; Dyslexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full Term children: born >36 weeks, currently age 6 +/- 6 months
- Preterm children: born <35 weeks, age 6 +/- 6 months at the beginning of the study.

SUMMARY:
The purpose of this study is to understand reading abilities of children born preterm: their cognitive profiles, the neural basis of good and poor reading abilities, and the behavioral and neural factors that predict persistent difficulties. The investigators hope to learn

* what specific skills correlate reading skills
* if preterm children have different cognitive profiles than full term children with respect to reading
* if cognitive skills measured in kindergarten predict reading ability in the second grade
* if parts of the brain are associated with reading skill
* whether brain characteristics in kindergarten predict reading in second grade.

DETAILED DESCRIPTION:
On the first day we will do the following:

1. We will ask your child to complete standardized tests of language, reading and intelligence.
2. We will ask you child to do computerized tests about grammar and higher mental functions, such as memory and planning.
3. While your child is doing tests, you will fill out some questionnaires and answer some questions about your child's health, behavior, and schooling. You may refuse to answer any individual question on the questionnaire.
4. We will review your child's medical records. Medical record review is for review of previous MRI scans and other conditions that might affect your child's ability in this study.

All participants will undergo the same cognitive and academic test battery initially at age 6 and again at age 8 years old.

On the day of the MRI scanning:

1. A member of the team will ask you and your child medical information to check that it is okay for your child to be tested.
2. Before your child begins the study, we will ask your child if s/he has had any medications, alcohol, tobacco, or over-the-counter drugs recently. If your child is taking stimulants for Attention-Deficit/Hyperactivity Disorder or ADHD (such as Ritalin, Concerta, Dexedrine, Adderall), antihistamines, pseudoephedrine or Sudafed, we will ask you to hold these medicines 24 hours before the scan. Your child can take them after the scan is complete. Deferring stimulants for 24 hours is safe and commonly done by many children with ADHD on weekends.
3. In the fMRI scanner, your child will lay on a table that slides inside the magnet. A technician will place your child's head in a head-coil (a helmet-like device) and make sure that s/he is comfortable. Your child will hold onto a ball that sounds an alarm when squeezed. This is a signal for the technician to stop the scan, come in to talk with your child, and take him or her out of the scanner if s/he is unable to continue with the tests. We will take pictures of the structure of your child's brain. During this time s/he can watch part of a video of his/her choice or one from our video library. In order for the brain pictures to come out right, it is very important that s/he does not move her/his head while inside the scanner. In between tasks, the technician will talk to your child through a microphone and ask if everything is OK. Your child should respond in a loud, clear voice without moving his/her head. We hope your child can complete the testing. Your child can choose to stop the testing at any time s/he needs to. Your child should tell the technician if anything is uncomfortable. You may sit in the scanning room if your child wants you to and if you don't have any metal in your body or any other MRI exclusions.

ELIGIBILITY:
Inclusion Criteria:

* Pre-terms: PT children born <35 weeks gestation and weighing <2000 grams at birth.
* Full-term: FT participants will be healthy children born ≥ 36 weeks gestation and weighing ≥ 2750 grams, who are developing typically per pediatrician well-visit report and match the PT group on age, gender, and SES.

Exclusion Criteria:

* Congenital anomalies or recognizable malformation syndromes
* Mother's self-reported use of illicit drugs or alcohol during pregnancy;
* Birth weight <3rd %tile (small for gestational age, SGA) according to gestational age specific growth curves;
* Serious neurological problems including active seizure disorder (afebrile seizure within the last year) and/or anticonvulsant medication use, history of a central nervous system infections, or ventriculoperitoneal shunt for treatment for hydrocephalus
* IQ < 70 on the testing of this study because we would expect language delays in this group;
* Sensori-neural hearing loss, defined as 4-tone pure-tone average > 25 decibels as assessed at any time because hearing loss compromises language and reading development;
* Visual impairments that would interfere with the ability to read; (8) presence of any other health condition that might compromise academic functioning (FT only).
* Any child who has not been learning English either at home or at school for at least 2 years

Ages: 57 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born <35 weeks (preterm) as compared to >36 weeks (full-term)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Feldman, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- See also: Stanford Center for Cognitive and Neurobiological Imaging — http://cni.stanford.edu/